CLINICAL TRIAL: NCT02399566
Title: Comparative Clinical Trial of Erlotinib and Pemetrexed for Maintenance Treatment in Lung Adenocarcinoma
Brief Title: Clinical Trial of Erlotinib and Pemetrexed for Maintenance Treatment in Lung Adenocarcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Jianhua Chen, MD, Hunan Province Tumor Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCTEBMTLA-2015
Record Dates: First submitted 2015-03-22; First posted 2015-03-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Lung Adenocarcinoma
Keywords: erlotinib; pemetrexed; maintenance therapy
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Erlotinib Hydrochloride; Pemetrexed

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): followed classical chemotherapy for 4 cycles, use Erlotinib orally for the maintenance therapy
  Interventions: Drug: Erlotinib, Pemetrexed
- Comparator (Active Comparator): followed classical chemotherapy for 4 cycles, use Pemetrexed interventional for the maintenance therapy
  Interventions: Drug: Erlotinib, Pemetrexed

INTERVENTIONS:
Drug: Erlotinib, Pemetrexed — followed classical chemotherapy for 4 cycles, use Erlotinib orally for the maintenance therapy.

SUMMARY:
The purpose of this study is to compare effects of erlotinib and pemetrexed as maintenance therapy for lung adenocarcinoma. Primary Outcome is the progression free survival (PFS). Based on prediction of different potential benefit groups, this study may help the oncologist to optimize and improve the maintenance therapy plan for lung adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically diagnosed stage III/IV Lung Adenocarcinoma;
* Age of 18-75years; Gender Not Required;
* Received systemic clinical examination, including chest X-ray, abdomen B ultrasound, head CT scan, radionuclide bone scan;
* Received cisplatin chemotherapy for 4 cycles before this study, the curative effect of chemotherapy is SD or above SD (efficacy evaluation time is 21 days, if it is SD, then the longest diameter of target lesions shall not increase);
* Adequate hematologic, renal, and hepatic function, Specific index as follows: liver function: S-Bilirubin ≤1.5 ULN ; Transaminase≤2 ULN. renal function: S-Creatinine ≤1.2 ULN; blood urea nitrogen ≤1.2 ULN . ULN: upper normal limit. Marrow Hemopoietic Function: WBC≥4.0×10^9/l, ANC≥2.0×10^9/l platelet count ≥100×10^9/l, Hb≥100 g/l;
* ECOG PS 0-2,Life expectancy ≥ 3 months; endure more than two cycle chemotherapy;
* The patients have explicit lung tumor lesions and the lesions were measurable; (According to the standard of RECIST1.1, they should have at least one of accurately measurable lesions with the largest diameter ≥ 10mm by spiral CT, MRI);
* No history of serious drug allergy;
* Informed consent should be obtained before treatment.

Exclusion Criteria:

* Not histologically or cytologically diagnosed as Lung Adenocarcinoma
* The age of >75 years or <18 years.
* Major organ dysfunction and Serious Heart Disease (congestive heart-failure, incontrollable high-risk arrhythmia, unstable angina, alular disease, myocardial infarct and Resistant hypertension,);
* Serious complications and investigator consider it is unsuited enrolling;
* Pregnant or lactating women;
* Allergic to research drug;
* Received cisplatin chemotherapy for 4 cycles before this study, the curative effect of chemotherapy is PD

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | two years

SECONDARY OUTCOMES:
Overall survival (OS) | two years
Clinical benefit rate (CBR) | two years
Objective response rate (ORR) | two years
The adverse reaction | two years
Time to progression (TTP) | two years